CLINICAL TRIAL: NCT04096508
Title: Application of Music Listening in Gastrointestinal Endoscopic Procedures
Brief Title: Role of Music Listening in Gastrointestinal Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 307-GIE-m
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Gastrointestinal Endoscopic Procedures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patients sit comfortably in a chair for 20 min listening classic music before the procedure.
  Interventions: Behavioral: Music listening
- Group B (Experimental): Patients sit comfortably in a chair for 20 min listening popular music before the procedure.
  Interventions: Behavioral: Music listening
- Control group (No Intervention): Patients sit comfortably in a chair for 20 min without music listening before the procedure.

INTERVENTIONS:
Behavioral: Music listening — Patients sit comfortably in a chair for 20 min listening music before the procedure.
  Arms: Group A; Group B

SUMMARY:
Gastrointestinal endoscopy is widely acknowledged as the most useful tool for diagnosing and treating gastrointestinal mucosal lesions. It can not only observe the mucosa directly, but also obtain tissue biopsy for pathological diagnosis. Although the importance of gastrointestinal endoscopy has been well understood, there are still a certain proportion of people who are unwilling to undergo it due to the discomfort and anxiety during the procedures. Music is multifunctional, which can alleviate people's depression, anxiety and other negative emotions as well as help to maintain good mental health. Thus, in this study we aim to investigate the role of music listening in gastrointestinal endoscopy in a randomized controlled clinical trial, especially for those patients who plan to undergo therapeutic endoscopic procedures and try to improve the patients' experience.

DETAILED DESCRIPTION:
This is a randomized controlled trial to examine the function of music listening in the procedures of gastrointestinal endoscopy. It was previously reported that music listening may exert beneficial effects for patients who undergo gastrointestinal endoscopy. However, most of the studies did not analyze the effects of the specific music type and listening time in diagnostic and therapeutic gastrointestinal endoscopic procedures, respectively. This study will test whether the specific music type and listening time before gastrointestinal endoscopy could improve patients' experience of the procedure in a randomized controlled trial. The results may help to optimize the routine clinical practice at present.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old patients
* Who agree to participate in the study
* Patients with the indications for gastrointestinal endoscopy

Exclusion Criteria:

* Patients, who were receiving nonsteroidal anti-inflammatory drugs, pump inhibitors (PPI) or antibiotics in the last 3 weeks.
* Severe uncontrolled coagulopathy
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | 4 months
  A 10-point scale was used to evaluate the patients' pain (0 least, 10 most). All the discomforts such as abdominal pain, distension and the like were all recorded.

SECONDARY OUTCOMES:
Patients' satisfaction and willingness to undergo gastrointestinal endoscopy again | 4 months
  A 10-point scale was used to evaluate the patients' satisfaction (0 worst, 10 best).
  It is anticipated that the use of music listening will significantly improve patients' satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee D, Henderson A, Shum D. The effect of music on preprocedure anxiety in Hong Kong Chinese day patients. J Clin Nurs. 2004 Mar;13(3):297-303. doi: 10.1046/j.1365-2702.2003.00888.x. PMID 15009332
- [Background] Hayes A, Buffum M, Lanier E, Rodahl E, Sasso C. A music intervention to reduce anxiety prior to gastrointestinal procedures. Gastroenterol Nurs. 2003 Jul-Aug;26(4):145-9. doi: 10.1097/00001610-200307000-00002. PMID 12920428
- [Background] Bechtold ML, Puli SR, Othman MO, Bartalos CR, Marshall JB, Roy PK. Effect of music on patients undergoing colonoscopy: a meta-analysis of randomized controlled trials. Dig Dis Sci. 2009 Jan;54(1):19-24. doi: 10.1007/s10620-008-0312-0. Epub 2008 May 16. PMID 18483858